CLINICAL TRIAL: NCT06169332
Title: Multidetector CT Left Appendage Atrial Thrombosis Exclusion in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: LATE
Record Dates: First submitted 2023-11-29; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Computed Tomography: Experimental computed tomography protocol: a few minutes after the administration of the contrast medium at a very low dose of radiation performed only in those patients in whom there is a doubt of thrombosis in the early arterial phase.

SUMMARY:
The aim of the LATE (multidetector CT Lefi Appendage atrial Thrombosis Exclusion in patients with atrial fibrillation) study is to evaluate the diagnostic accuracy of cardiac Computed Tomography (TC) with 64 detectors and double acquisition phase in candidate patients ablation of atrial fibrillation (AF) with the Navx (or Carto) technique, using trans-esophageal ultrasound (TEE) as the standard reference.

This study is based on the use of an experimental protocol in cardiac TC which involves, in addition to the acquisition of an early arterial phase (standard protocol routinely performed in all patients), the execution of a possible late phase at a very low dose of radiation (experimental protocol) aimed at increasing the accuracy of the method in the diagnosis in patients with AF. The LATE study aims to demonstrate the high diagnostic accuracy of dual acquisition phase cardiac TC in the diagnosis of intraauricular thrombosis by comparing it with reference standard; in light of this result, cardiac TC could constitute a single non-invasive diagnostic tool in the future for the global evaluation of both atrial anatomy and endoawicular thrombosis with a clear improvement in patient management both in clinical and economic terms.

ELIGIBILITY:
Inclusion Criteria:

* patients candidates for cardiac TC and transesophageal ultrasound examination for the evaluation of cardiac anatomy and for the exclusion of intra-auricular thrombosis.

Exclusion Criteria:

* < 18 years patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom there is a doubt of thrombosis in the early arterial phase.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2013-03-25 (Actual)

PRIMARY OUTCOMES:
Cardiac computed tomography for the staging of patients with intraauricular thrombosis. | 3 years
  evaluation of the diagnostic accuracy of cardio CT in the diagnosis of intraauricular thrombosis in patients candidates for atrial fibrillation ablation.